CLINICAL TRIAL: NCT02410395
Title: NIche Development With Closure of Cesarean Uterotomy by Modified or Conventional Two-layer Technique (NICUM Study)
Brief Title: NIche Development With Closure of Cesarean Uterotomy by Modified or Conventional Two-layer Technique
Acronym: NICUM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AUH060804
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Cesarean Scar Niche
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional technique (Active Comparator): Closure of the uterotomy with a conventional two-layer technique
  Interventions: Procedure: Conventional
- Modified technique (Experimental): Closure of the uterotomy with a modified two-layer technique
  Interventions: Procedure: Modified

INTERVENTIONS:
Procedure: Conventional — Two-layer technique with the first layer performed as an un-locked, continuous suture without inclusion of the endometrium and the second layer performed as an un-locked, continuous suture with the stitches placed superficially, horizontally along the first layer.
  Arms: Conventional technique
Procedure: Modified — The modified mattress suture is performed as a single-suture, double-layer technique with limited inclusion of the myometrium and broad inclusion of the serosal surface and myometrium, interchangeably
  Arms: Modified technique

SUMMARY:
The aim of this trial was to compare two different uterotomy surgical techniques on the occurrence of a uterine niche and the risk of a number of short- and long-term gynecological complications associated with the presence and size of the niche.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnant
* Intended elective cesarean section

Exclusion Criteria:

* Cervical dilatation of more than 4 cm
* Previous cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Presence of a cesarean scar niche more than 2 mm deep. | 6 months

SECONDARY OUTCOMES:
Residual myometrial thickness of the cesarean scar (RMT) | 6 months
Cesarean scar niche depth, width, length, myometrium adjacent to the scar | 6 months
Post-menstrual spotting | 15 months
Incidence of cesarean scar pregnancy or spontaneous abortions | 72 months
Adverse pregnancy outcomes in the following pregnancy | 72 months
  Composite of placenta previa, placenta accreta or percreta, uterine rupture or dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Niels Uldbjerg, MD, DMSc, Study Chair — Aarhus University Hospital; Lone Hvidman, MD, PhD, Study Chair — Aarhus University Hospital; Axel Forman, MD, DMSc, Study Chair — Aarhus University Hospital
Locations (1):
- Dep. Obstetrics and Gynecology, Regional Hospital of Randers, Randers, Denmark